CLINICAL TRIAL: NCT02936674
Title: Color-dependent Melatonin Suppression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jamie M. Zeitzer, Ph.D., Assistant Professor, VA Palo Alto Health Care System
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRB-10165
Record Dates: First submitted 2016-10-07; First posted 2016-10-18 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Light 1 (Experimental): Light 1 will have an altered color composition as compared with a standard LED bulb.
  Interventions: Device: Light - alternate
- Light 2 (Active Comparator): Light 2 will be a standard LED bulb.
  Interventions: Device: Light - standard

INTERVENTIONS:
Device: Light - standard — Light will be given during the night to determine its effects on melatonin suppression. This light will be an LED with standard spectral distribution
  Arms: Light 2
Device: Light - alternate — Light will be given during the night to determine its effects on melatonin suppression. This light will be an LED with an altered spectral distribution (different color)
  Arms: Light 1

SUMMARY:
The purpose of this study is to examine the effects of complex, broad-band spectra light on the production of melatonin in humans.

ELIGIBILITY:
Inclusion Criteria:

* Stable health
* Normal color vision
* Normal hearing
* 18-35 years old

Exclusion Criteria:

* Significant depressive symptoms
* Pregnant or nursing
* Ocular pathologies
* Unstable or severe medical or psychiatric condition
* Extreme morning/evening type
* Regular smoker
* Use of medications that impact ocular function
* Alcohol use disorder
* Use of illegal drugs
* Irregular use of antihistamines, antidepressants, or sleeping medications

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-10; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Melatonin suppression | 4 Hours
  The amount of declination of salivary melatonin concentrations between the start of the light and the end of the light (4 hours later) will be compared between the conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All relevant individual data will be published.